CLINICAL TRIAL: NCT02654808
Title: A Comparison of CO2 Absorption During Gynecologic Laparoscopy Using the AirSeal® Valveless Trocar System Versus Standard Insufflation Trocars at Intra-abdominal Pressures of 10 mmHg and 15 mmHg - a Randomized Controlled Trial
Brief Title: AirSeal®Insufflation Trocar/CO2 Absorption Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAQ6474
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Gynecologic Diseases
Keywords: Gynecology; Laparoscopy; Pneumoperitoneum; CO2 absorption
MeSH Terms: conditions — Genital Diseases, Female; Pneumoperitoneum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Standard trocar/ IAP 15 mmHg (Active Comparator): Patients who are randomized into this arm will have their laparoscopic procedures performed with the standard trocar insufflator at an intra-abdominal pressure (IAP) of 15 mmHg.
  Interventions: Device: Standard trocar
- Standard trocar/ IAP 10 mmHg (Active Comparator): Patients who are randomized into this arm will have their laparoscopic procedures performed with the standard trocar insufflator at an intra-abdominal pressure (IAP) of 10 mmHg.
  Interventions: Device: Standard trocar
- AirSeal trocar/ IAP 15 mmHg (Active Comparator): Patients who are randomized into this arm will have their laparoscopic procedures performed with the AirSeal trocar insufflator at an intra-abdominal pressure (IAP) of 15 mmHg.
  Interventions: Device: AirSeal trocar
- AirSeal trocar/ IAP 10 mmHg (Active Comparator): Patients who are randomized into this arm will have their laparoscopic procedures performed with the AirSeal trocar insufflator at an intra-abdominal pressure (IAP) of 10 mmHg.
  Interventions: Device: AirSeal trocar

INTERVENTIONS:
Device: AirSeal trocar — The AirSeal® trocar is a valveless trocar that has been designed to replace the "trap door" and silicone valve of standard trocars with a curtain of forced CO2 gas. With the AirSeal® trocar, escaping gas is collected at the proximal end of the trocar, filtered, and redirected into the peritoneal cavity to maintain the pressure differential. The result is an invisible barrier that instantaneously responds to changes in intra-abdominal pressure, either by allowing more CO2 inflow with pressure drops or by serving as a pressure relief valve during pressure spikes.
  Arms: AirSeal trocar/ IAP 10 mmHg; AirSeal trocar/ IAP 15 mmHg
Device: Standard trocar — A standard insufflation trocar delivers CO2 into the abdominal cavity to create workspace and uses either a "trap door" or silicone valve to prevent the egress of CO2 during laparoscopy in order to maintain intra-abdominal pressures. The standard trocars are not equipped to respond to changes in the intra-abdominal pressures in order to trigger an increase or decrease in the flow rate of CO2 gas.
  Arms: Standard trocar/ IAP 10 mmHg; Standard trocar/ IAP 15 mmHg

SUMMARY:
The purpose of this study is to compare carbon dioxide (CO2) absorption during gynecologic laparoscopy using the AirSeal® valveless trocar system versus standard insufflation trocars at intra-abdominal pressures of 10 and 15 mmHg.

The investigators hypothesize that with the AirSeal® valveless trocar system, gynecologic laparoscopy can be performed at a lower intra-abdominal pressure with a possible resultant decrease in CO2 absorption, while maintaining adequate visualization of the operative field for safe completion of surgery.

DETAILED DESCRIPTION:
Three main factors affect patients' cardiopulmonary status during gynecologic laparoscopy: 1) degree of Trendelenburg tilt (25 - 30°), 2) carbon dioxide (CO2) absorption and 3) increased intra-abdominal pressure (10 -20 mmHg). Slight modifications to any or all of these three factors can lead to a significant decrease in morbidity.

The AirSeal® valveless trocar system reduces CO2 absorption when compared to standard trocars during renal laparoscopy. Also, use of this trocar system provides a more stable intra-abdominal pressure when compared to standard trocars, a feature that could possibly allow for laparoscopic surgery to be performed at lower intra-abdominal pressures.

ELIGIBILITY:
Inclusion Criteria:

* Any woman ≥ 18 years of age undergoing a gynecologic laparoscopic procedure
* Able to understand the consenting process and willing to participate in study

Exclusion Criteria:

* Patient unable to undergo laparoscopic procedure due to size of pathology or medical comorbidities
* Emergent surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ryntz, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herati AS, Andonian S, Rais-Bahrami S, Atalla MA, Srinivasan AK, Richstone L, Kavoussi LR. Use of the valveless trocar system reduces carbon dioxide absorption during laparoscopy when compared with standard trocars. Urology. 2011 May;77(5):1126-32. doi: 10.1016/j.urology.2010.06.052. Epub 2010 Oct 2. PMID 20888033
- [Background] Tan PL, Lee TL, Tweed WA. Carbon dioxide absorption and gas exchange during pelvic laparoscopy. Can J Anaesth. 1992 Sep;39(7):677-81. doi: 10.1007/BF03008229. PMID 1394755
- [Background] Gerges FJ, Kanazi GE, Jabbour-Khoury SI. Anesthesia for laparoscopy: a review. J Clin Anesth. 2006 Feb;18(1):67-78. doi: 10.1016/j.jclinane.2005.01.013. PMID 16517337
- [Background] Rauh R, Hemmerling TM, Rist M, Jacobi KE. Influence of pneumoperitoneum and patient positioning on respiratory system compliance. J Clin Anesth. 2001 Aug;13(5):361-5. doi: 10.1016/s0952-8180(01)00286-0. PMID 11498317
- [Background] CONMED - Transforming Laparosopic Surgery. Available at: http://www.conmed.com/en/hybrid-product-landing-pages/airseal. Retrieved January 12, 2018.
- [Background] Wolf JS Jr, Monk TG, McDougall EM, McClennan BL, Clayman RV. The extraperitoneal approach and subcutaneous emphysema are associated with greater absorption of carbon dioxide during laparoscopic renal surgery. J Urol. 1995 Sep;154(3):959-63. PMID 7637101
- [Background] Ng CS, Gill IS, Sung GT, Whalley DG, Graham R, Schweizer D. Retroperitoneoscopic surgery is not associated with increased carbon dioxide absorption. J Urol. 1999 Oct;162(4):1268-72. PMID 10492177
- [Background] Motew M, Ivankovich AD, Bieniarz J, Albrecht RF, Zahed B, Scommegna A. Cardiovascular effects and acid-base and blood gas changes during laparoscopy. Am J Obstet Gynecol. 1973 Apr 1;115(7):1002-12. doi: 10.1016/0002-9378(73)90683-2. No abstract available. PMID 4266615
- [Background] Joshipura VP, Haribhakti SP, Patel NR, Naik RP, Soni HN, Patel B, Bhavsar MS, Narwaria MB, Thakker R. A prospective randomized, controlled study comparing low pressure versus high pressure pneumoperitoneum during laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2009 Jun;19(3):234-40. doi: 10.1097/SLE.0b013e3181a97012. PMID 19542853
- [Background] Sefr R, Puszkailer K, Jagos F. Randomized trial of different intraabdominal pressures and acid-base balance alterations during laparoscopic cholecystectomy. Surg Endosc. 2003 Jun;17(6):947-50. doi: 10.1007/s00464-002-9046-9. Epub 2003 Mar 14. PMID 12632130
- [Background] Vijayaraghavan N, Sistla SC, Kundra P, Ananthanarayan PH, Karthikeyan VS, Ali SM, Sasi SP, Vikram K. Comparison of standard-pressure and low-pressure pneumoperitoneum in laparoscopic cholecystectomy: a double blinded randomized controlled study. Surg Laparosc Endosc Percutan Tech. 2014 Apr;24(2):127-33. doi: 10.1097/SLE.0b013e3182937980. PMID 24686347
- [Background] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Background] Park JS, Ahn EJ, Ko DD, Kang H, Shin HY, Baek CH, Jung YH, Woo YC, Kim JY, Koo GH. Effects of pneumoperitoneal pressure and position changes on respiratory mechanics during laparoscopic colectomy. Korean J Anesthesiol. 2012 Nov;63(5):419-24. doi: 10.4097/kjae.2012.63.5.419. Epub 2012 Nov 16. PMID 23198035
- [Background] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939
- [Background] Kandil TS, El Hefnawy E. Shoulder pain following laparoscopic cholecystectomy: factors affecting the incidence and severity. J Laparoendosc Adv Surg Tech A. 2010 Oct;20(8):677-82. doi: 10.1089/lap.2010.0112. PMID 20701547
- [Background] Bogani G, Uccella S, Cromi A, Serati M, Casarin J, Pinelli C, Ghezzi F. Low vs standard pneumoperitoneum pressure during laparoscopic hysterectomy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):466-71. doi: 10.1016/j.jmig.2013.12.091. Epub 2013 Dec 25. PMID 24374246

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Trocar/ IAP 15 mmHg | Standard Trocar/ IAP 10 mmHg | AirSeal Trocar/ IAP 15 mmHg | AirSeal Trocar/ IAP 10 mmHg
Started | 33 | 33 | 33 | 33
Completed | 33 | 33 | 33 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Trocar/ IAP 15 mmHg | Standard Trocar/ IAP 10 mmHg | AirSeal Trocar/ IAP 15 mmHg | AirSeal Trocar/ IAP 10 mmHg | Total
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 33 | 33 | 132
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 33 | 33 | 132
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 9 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 9 | 13 | 8 | 4 | 34
  White | 14 | 12 | 6 | 17 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 10 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Average Carbon Dioxide (CO2) Absorption During Gynecologic Laparoscopy Using the AirSeal® Versus Standard Trocars at Intra-abdominal Pressures of 10 mmHg
Description: This outcome is measured by calculating the CO2 elimination rate. CO2 absorption rates were obtained at 15 and 60 minutes during each case and an average value was calculated per case. In cases < 60 minutes, the CO2 absorption rate at 15 minutes will be used.
Time Frame: 15 minutes & 60 minutes from surgery start time
Population: 132 patients were enrolled and randomized into 1 of 4 study arms: standard insufflation/IAP 10 (S/10), standard insufflation/IAP 15 (S/15), valveless insufflation/IAP 10 (V/10), valveless insufflation/IAP 15 (V/15).
Measure: Mean (Standard Deviation); unit: mL/(kg*min)
Arm/Group | Standard Trocar/ IAP 15 mmHg | Standard Trocar/ IAP 10 mmHg | AirSeal Trocar/ IAP 15 mmHg | AirSeal Trocar/ IAP 10 mmHg
Number analyzed (Participants) | 31 | 32 | 32 | 33
mL/(kg*min) | 3.96 (1.19) | 4.05 (1.08) | 4.04 (1.54) | 3.97 (1.00)

2. Secondary Outcome: Median Surgeon Questionnaire Score When Using AirSeal® Versus Standard Trocars
Description: Surgeon Questionnaire (0 "not adequate" -10 "optimal") is designed to evaluate the visualization of operative field by surgeon during colpotomy.
Time Frame: At the end of surgery (approximately 1 hour)
Population: 132 patients were enrolled and randomized with 33 patients per arm. The participants were women ≥ 18 years old undergoing non-emergent conventional or robotic gynecologic laparoscopic surgery.
Measure: Median (Standard Deviation); unit: score on a scale from 0 to 10
Groups:
- Standard 10: Standard insufflation system 10mmHg
- Standard 15: standard insufflation system 15 mmHg
- Valveless 10: Valveless insufflation system 10 mmHg
- Valveless 15: Valveless insufflation system 15 mmHg
Arm/Group | Standard 10 | Standard 15 | Valveless 10 | Valveless 15
Number analyzed (Participants) | 32 | 31 | 33 | 32
score on a scale from 0 to 10
  Baseline | 10.0 (2.0) | 10.0 (1.0) | 10.0 (1.0) | 10.0 (0.8)
  At 15 minutes | 8.0 (3.0) | 8.0 (4.0) | 10.0 (2.0) | 10.0 (2.0)
  At 30 minutes | 8.0 (3.0) | 8.0 (3.0) | 9.0 (3.0) | 9.0 (2.0)
  Colpotomy | 4.5 (4.0) | 5.0 (4.0) | 8.0 (4.0) | 9.0 (2.0)
  Overall | 7.0 (3.0) | 7.0 (2.0) | 9.0 (2.0) | 9.5 (1.8)

3. Secondary Outcome: Number of Participants With no Problem When Using AirSeal® Versus Standard Trocars
Description: Anesthesia Questionnaire (0 "no problem" - 2 "very problematic) is designed to evaluate the the level of difficulty in maintaining adequate end-tidal CO2 (etCO2).
Time Frame: At the end of surgery (approximately 1 hour)
Population: Women ≥ 18 years old undergoing non-emergent conventional or robotic gynecologic laparoscopic surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 10 | Standard 15 | Valveless 10 | Valveless 15
Number analyzed (Participants) | 32 | 31 | 33 | 32
Participants | 30 | 30 | 32 | 32

4. Secondary Outcome: Median VAS Pain Score When Using AirSeal® Versus Standard Trocars
Description: Visual Analog Scale (VAS) Pain Score (0 "no pain" - 10 "worst pain") is designed to evaluate the level of pain post-surgery.
Time Frame: 4 to 6 hours, and 12 to 23 hours following surgery
Population: Post-operative shoulder pain of women ≥ 18 years old undergoing non-emergent conventional or robotic gynecologic laparoscopic surgery.
Measure: Median (Standard Deviation); unit: score on a scale from 0 to 10
Arm/Group | Standard 10 | Standard 15 | Valveless 10 | Valveless 15
Number analyzed (Participants) | 32 | 31 | 33 | 32
score on a scale from 0 to 10
  PACU arrival | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  PACU discharge | 0 (2) | 0 (0) | 0 (4) | 0 (1)
  Post-operative Day #1 | 0 (4) | 0 (4) | 0 (4) | 0 (5)
  4 to 6 hours | 0 (5) | 0 (0) | 0 (0) | 0 (9)
  12 to 23 hours | 0 (0) | 0 (0) | 0 (2) | 1.5 (7)

5. Secondary Outcome: Average Carbon Dioxide (CO2) Absorption During Gynecologic Laparoscopy Using the AirSeal® Versus Standard Trocars at Intra-abdominal Pressures of 15 mmHg
Description: This outcome is measured by calculating the CO2 elimination rate.
Time Frame: 15 minutes & 60 minutes from surgery start time
Population: Women ≥ 18 years old undergoing non-emergent conventional or robotic gynecologic laparoscopic surgery.
Measure: Mean (Standard Deviation); unit: mL/(kg*min)
Arm/Group | Standard 10 | Standard 15 | Valveless 10 | Valveless 15
Number analyzed (Participants) | 32 | 31 | 33 | 32
mL/(kg*min) | 4.05 (1.08) | 3.96 (1.19) | 3.97 (1.00) | 4.04 (1.54)

ADVERSE EVENTS:
Time Frame: Up to 1 day following surgery
Arm/Group | Standard Trocar/ IAP 15 mmHg | Standard Trocar/ IAP 10 mmHg | AirSeal Trocar/ IAP 15 mmHg | AirSeal Trocar/ IAP 10 mmHg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02654808/Prot_SAP_000.pdf